CLINICAL TRIAL: NCT06305026
Title: Diagnostic Test Accuracy of Histological Muscle and Skin Biopsies of Rheumatoid Arthritis Patients Revealing Objective Chronic Widespread Pain Phenomena Related to Fibromyalgia
Brief Title: Protocol for a Diagnostic Test Accuracy of Histological Muscle and Skin Biopsies of Rheumatoid Arthritis Patients Revealing Objective Chronic Widespread Pain Phenomena Related to Fibromyalgia
Status: Completed | Type: Observational
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Philip Rask Lage-Hansen, MD, Esbjerg Hospital - University Hospital of Southern Denmark
Other Study IDs: S-20190160
Record Dates: First submitted 2024-02-22; First posted 2024-03-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis; Fibromyalgia, Secondary; Widespread Chronic Pain; Muscle Disorder
MeSH Terms: conditions — Arthritis, Rheumatoid; Fibromyalgia; Chronic Pain; Muscular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Muscle Biopsies and skin biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RA patients with concomitant fibromyalgia
  Interventions: Diagnostic Test: Muscle- and skin biopsies
- RA patients without concomitant fibromyalgia
  Interventions: Diagnostic Test: Muscle- and skin biopsies

INTERVENTIONS:
Diagnostic Test: Muscle- and skin biopsies — RA patients with and without concomitant fibromyalgia will be examined with muscle and skin biopsies.

SUMMARY:
Background: Chronic widespread pain is challenging in the management of the patient with rheumatoid arthritis (RA), affecting approximately one third of this patient population. However, pain is not always caused by disease activity (inflammation) but can be associated to central pain mechanisms as seen in fibromyalgia (FM). FM is characterized by widespread pain and tenderness; often accompanied by disturbed sleep, fatigue, cognitive impairment, emotional distress and multiple symptoms from various organ systems. Among patients with RA the prevalence of concomitant FM is reported to be 12-17% compared to 1-3% in the general population. In general the pain, felt by the fibromyalgia patients is considered to be due to lower pain thresholds because of abnormal central pain processing. Pain reported by RA patients with concomitant FM could potentially be explained by this phenomenon. Little is known about RA patients fulfilling criteria for FM. Muscles-studies of FM patients have not found any histopathological explanation of the pain felt, however an old study of muscle changes in RA patients found changes that could explain muscle pain. Small fiber neuropathy (SFN) is a condition associated with autoimmune diseases, and evidence suggests that SFN is likely to contribute to the pain observed in FM.

Objectives: To determine the diagnostic test accuracy (sensitivity and specificity) of both muscle- and skin-biopsies for fibromyalgia phenotyping and detection by clinical referral (RA with concomitant FM) as the reference standard (i.e. fulfilment of 2016 FM criteria).

Data collection: Will be done as study subjects are included and stored in REDCAP.

Eligibility criteria for participants and settings where the data will be collected: RA patients will be assessed in the daily clinic in Esbjerg and Odense and examined for concomitant FM (I.e. satisfying the 2016 criteria for FM). Patients will afterwards be invited to participate in the study. Inclusion will continue until 25 RA patients fulfilling FM criteria and thus based on the expected prevalence at least 25 (- and maximum 50) RA patients not fulfilling FM critieria has undergone the index tests.

Whether participants form a consecutive, random, or convenience series: Participants form a consecutive series.

Description of the index test and reference standard: Twenty-five RA patients with concomitant FM and more than 25 (- maximum 50 patients) RA patients not fulfilling FM criteria will undergo the index tests. Muscle and skin biopsies will be performed in each group using standardized techniques. The reference standard will be fulfillment of the 2016 criteria for fibromyalgia.

Estimates of diagnostic accuracy and their precision: Regarding muscle- and skin biopsies sensitivity, specificity and positive predictive value will be calculated using two times two table. Regarding skin biopsies, median values in the two groups (RA +/- FM) will be compared using a two-sample t-test.

DETAILED DESCRIPTION:
To determine the diagnostic test accuracy (the sensitivity and specificity) of both muscle- and skin-biopsies for fibromyalgia phenotyping and detection by clinical referral (RA with concomitant CWP) as the reference standard (i.e. fulfilment of 2016 FM criteria).

Background Pain poses a huge challenge in the management of Rheumatoid arthritis (RA) patients, affecting approximately half of this patient population, even in patients with low disease activity. 1/3 report significant pain. As the composite DAS-28 score has become the standard tool for monitoring RA patients in daily routine, the patient's history of joint pain is of great importance as it influences the VAS applied for patient global assessment and the tender joint count (TJC), which is the single factor with the highest impact on the final DAS-28 score. However, the TJC score is not always associated with clinically quantified inflammation but can be associated with central pain mechanisms, as seen in Fibromyalgia (FM). FM is characterized by widespread pain and tenderness, often accompanied by disturbed sleep, fatigue, cognitive impairment, emotional distress, and multiple symptoms from various organ systems. The prevalence of FM varies between 1-3 percent in the general population. However, among patients with RA, the prevalence is reported to be 12-17%.

The sensation of pain is a product of the interaction of multiple processes. Nociceptors transduce mechanical, chemical, or thermal stimuli into electric signals, which are transmitted through the dorsal horn of the spinal cord to the brainstem and higher cortical areas. The Periaqueductal grey substance (PAG) and the rostral ventromedial medulla (RVM) modulate the pain signal through descending pathways to the dorsal horn of the medulla. In chronic pain states, changes in nociceptive signaling may involve sensitization of nociceptive neurons and ascending spinal tracts accompanied by dysfunction of descending pain modulatory pathways. Changes in nociceptive signaling with lowering of pain thresholds could be an explanation of a high TJC in RA patients if inflammation is not present. As RA patients with FM have similar complaints to patients with primary FM, including former histopathology studies in FM is relevant. Several muscle biopsy studies have been performed on FM patients with conflicting results. Four studies found no differences, three studies report changes associated with ischemia, and few studies report differences between muscle biopsies obtained from FM and healthy controls; however, no pathognomonic pathology in the FM muscles has been detected. Today, consensus exists regarding pathology in muscle biopsies with inflammatory myopathy, which was not the case when all earlier studies were performed. In our study, we apply this method to muscle biopsies from patients with RA and fibromyalgia.

Polyneuropathy is associated with autoimmune diseases. Evidence suggests that small fiber neuropathy (SFN) is likely to contribute to the pain in FM. In skin biopsies, SFN is associated with intra-epidermal nerve fiber density (IENFD). It can be evaluated histologically and quantified. The technique has recently been validated. No muscle or skin biopsy study has been performed on RA patients with or without concomitant FM.

Research question and aim. To determine the sensitivity and specificity of both muscle- and skin biopsies for fibromyalgia phenotyping and detection by clinical referral (RA with concomitant CWP) as the reference standard (i.e., fulfillment of 2016 FM criteria).

Hypotheses

1. Muscle biopsies from RA patients with concomitant FM are histologically different compared to RA patients without FM.
2. Skin biopsies from RA patients with concomitant FM are histologically different regarding the quantitative histological evaluation of intraepidermal nerve fiber (IENF) density compared to RA patients without FM.

METHODS Methods: RA patients with FM will be consecutively invited during their regular visits to the outpatient clinics of Rheumatology in Esbjerg and Odense. When signed consent has been given, patients will be examined for the fulfillment of criteria for concomitant fibromyalgia. If satisfying the inclusion criteria (and absence of exclusion criteria (see below)), they will undergo muscle and skin biopsy and blood sampling. Study participants recruited will all be characterized clinically by anti-citrullinated protein antibody and Immunoglobulin M rheumatoid factor (ACPA/IgM-RF) status, D-vitamin and Creatin kinases (CK) level and myositis antibodies in the blood, tender- and swollen joint counts (TJC and SJC), Health assessment questionnaire disability index status (HAQ-status) and acute phase reactant (CRP) will be measured. Moreover, patients' evaluation of pain and fatigue, a global assessment by visual analog scales (VAS), tender point evaluation (TP), and examination for the fulfillment of the 1990 ACR criteria for FM and the 2016 criteria for FM will be noted.

Furthermore, the cold pressor test, pain pressure threshold (PPT) over m. masseter and computerized cuff pressure algometry (CPA) will be performed in all patients (see below). The clinical evaluation and characterization of immunology status and pain measurements are performed before muscle and skin biopsies. Enrolment will be done consecutively until 25 RA patients fulfill FM criteria, and thus, at least 25 (- maximum 50 patients) not fulfilling the criteria for FM are met.

Pain test Pain test: Three different pain tests are performed in order to characterize the pain tolerance and pain threshold, which is assumed to be lower in RA patients with concomitant fibromyalgia.

Cold pressure test: In this test, the hand is immersed into water with a temperature of 1-6 degrees Celsius. Two main measures are derived: Pain threshold is defined as the time when the subject indicates noticeable pain and pain tolerance is defined as the elapsed time from exposure to cold water to the point where the subject withdraws the hand from the water because of the pain felt.

Pain pressure threshold (PPT): In this test, an increasing pressure is applied to the muscle in the jaw. The pressure applied until the subject indicates noticeable pain defines pain threshold.

Computerized Cuff pressure algometry (CPA): Pressure pain sensitivity is determined on the lower leg. The setup includes a pneumatic tourniquet cuff, a computerized compressor, and an electronic 10 cm Visual Analogue Scale (VAS). Double-chambered textile TourniquetCuffs (VBM Medizintechnik GmbH, Sulz, Germany) are applied for pressure. Measurements are carried out with the patient in the supine position and on the patient's dominant side. At all measurements a compression rate of 1.0kPa/sec is used. To minimize bias due to the summation of pain, all measurements are carried out with a time interval of 5 minutes (the stimulus is repeated three times). Pain Threshold is defined as the pressure of the cuff at the subject's first sensation of pain when applying a constantly rising pressure (Unit kPa). Pain tolerance is defined as the pressure of the cuff when the patient switches off the pressure due to worst tolerable pain caused by pressure stimulation (Unit kPa).

Eligibility criteria: Patients with known RA satisfying the 2010 criteria for RA.

Inclusion criteria Age equal to or over 18. RA patient.

Exclusion criteria Alcohol abuse, wheelchair users, and patients who require personal assistance with daily activities. Medication with glucocorticoids within the last 6 weeks. A diagnosis of a systemic autoimmune disease other than RA, peripheral vascular disease manifested by claudication or ischemic rest pain, neuropathy, and diabetes. Patients with abnormal TSH levels.

Biopsies

1. Five mm long and 3 mm width incision biopsies of skeletal muscle will be evaluated by microscopy regarding inflammation, signs of neurogenic involvement, signs of dystrophy, and myopathy. The proportion of patients in each group (RA with and without FM) will be compared regarding muscle fibers, the vascular domain, connective tissue, and inflammation. A muscle pathologist will evaluate the muscle biopsies and is blinded to all clinical information.
2. 3 mm punch skin biopsies will be evaluated regarding IENFD density. The proportion of patients in each group (RA with and without FM) will be compared. The investigator evaluating the skin biopsies is blinded to all clinical information.

Index test: Two different tests will be examined regarding their ability to identify RA patients with concomitant fibromyalgia.

Index test #1 (Muscle biopsy): Two biopsies from every patient will be necessary. The proportion of patients in each group (RA with and without FM) will be compared regarding: muscle fibers, the vascular domain, connective tissue and inflammation (non-parametric test's). International consensus exists regarding clear histological signs of disease and therefore dichotomization is feasible and relevant.

Index test #2 (Skin biopsy): 3 mm punch skin biopsies 10 cm proximal from the right ankle will be evaluated regarding IENFD density. The proportion of patients in each group (RA with and without FM) will be compared (non-parametric test).

Definition of and rationale for test #1 (Muscle biopsy) positivity cut-offs: The muscle pathologists evaluate the muscle biopsies, and test results will be reported as dichotomous, pathological, or non-pathological according to international consensus.

Definition of and rationale for test #2 (Skin biopsy) positivity cut-offs: Skin biopsies will be evaluated regarding intra epidermal nerve fiber density (IENFD). The scale is continuous, and median values in the two groups (RA +/- FM) will be compared. IENFD will be considered abnormal according to values outside the 95% percentile of the normal range.

Definition of and rationale for reference standard positivity cut-offs: The reference standard is the fulfillment of the 2016 criteria for FM. The cut offs are dichotomous. Either patients fulfill the criteria, or they do not.

Training and expertise of the persons executing and reading the tests:

Two highly experienced muscle pathologists will evaluate the muscle biopsies and be blinded to all clinical information. Two experienced rheumatologists will be performing the muscle- and skin biopsies. The investigator evaluating the skin biopsies is blinded to all clinical information and is highly experienced in the field.

Statistical Methods Power and sample size considerations: No other study has been performed in this patient group earlier, so no formal power calculation could be done. Muscle pathologists were asked how many biopsies they thought necessary, and 25 in the RA-FM group was considered enough (and still feasible). Estimation and comparison of diagnostic accuracy: Regarding muscle biopsies, sensitivity, specificity, and positive predictive value will be calculated using two times two tables.

Regarding skin biopsies, median values in the two groups (RA +/- FM) will be compared, and an unpaired t-test will be applied for statistical calculation. P-value < 0.05 will be considered significant. Values deviating from the 95 percentiles according to age and gender regarding IENFD are defined as abnormal. Sensitivity, specificity, and positive predictive value will be calculated using two times two tables.

Handling of indeterminate index test or reference standard results: The muscle biopsies test results are dichotomous. Both muscle pathologists will evaluate indeterminate results and make a consensus. The final result will be pathologically yes/no. The skin biopsies measure intra-epidermal nerve fiber density (IENFD). The scale is continuous, and the median values of the two groups (RA +/- FM) will be compared. Cut of value separates normal from abnormal; no indeterminate test result will be possible.

Handling missing data on the index test and reference standard: Patients will be excluded from the study if the index is not performed.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or over 18
* RA patient

Exclusion Criteria:

* Alcohol abuse
* Wheelchair users, and patients who require personal assistance with daily activities.
* Medication with glucocorticoids within the last 6 weeks.
* A diagnosis of a systemic autoimmune disease other than RA
* Peripheral vascular disease manifested by claudication or ischemic rest pain
* Neuropathy
* Diabetes
* Patients with abnormal TSH levels.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: RA patients with or without concomitant fibromyalgia
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Muscle pathology | The biopsies will be performed the day the patients give written consent coresponding to day/time of inclusion. Estimated period of time over which the event is assessed is 40 weeks.
  Two muscle biopsies from every patient will be necessary. The proportion of patients in each group (RA with and without FM) will be compared regarding muscle fibers, the vascular domain, connective tissue, and inflammation (non-parametric tests). International consensus exists regarding clear histological signs of disease; therefore, dichotomization is feasible and relevant. Definition of and rationale for test #1 (Muscle biopsy) positivity cut-offs: The muscle pathologists evaluate the muscle biopsies, and the test result will be reported as dichotomous, that is, pathological or non-pathological according to international consensus.
Skin biopsies | The biopsies will be performed the day the patients give written consent coresponding to day/time of inclusion. Estimated period of time over which the event is assessed is 40 weeks.
  3 mm punch skin biopsies 10 cm proximal from the right ankle will be evaluated regarding IENFD density. The proportion of patients in each group (RA with and without FM) will be compared (non-parametric test). Definition of and rationale for test #2 (Skin biopsy) positivity cut-offs: Skin biopsies regarding intra epidermal nerve fiber density (IENFD) will be evaluated. IENFD will be considered abnormal according to values outside the 95% percentile of the normal range according to age. The proportion of patients with abnormal values will be compared in the two groups.

SECONDARY OUTCOMES:
Cold pressure test | The Test will be performed the day the patients give written consent coresponding to day/time of inclusion. Estimated period of time over which the event is assessed is 40 weeks.
  In this test, the hand is immersed in water at 1-6 degrees Celsius. Two main measures are derived: Pain threshold, defined as the time when the subject indicates noticeable pain, and pain tolerance, defined as the elapsed time from exposure to cold water to the point where the subject withdraws the hand from the water because of the pain felt.
Pain pressure threshold (PPT) | The Test will be performed the day the patients give written consent coresponding to day/time of inclusion. Estimated period of time over which the event is assessed is 40 weeks.
  In this test, an increasing pressure is applied to the muscle in the jaw. The pressure applied (measured in kg) until the subject indicates noticeable pain defines pain threshold.
Computerized Cuff pressure algometry (CPA) | The Test will be performed the day the patients give written consent coresponding to day/time of inclusion. Estimated period of time over which the event is assessed is 40 weeks.
  Pressure pain sensitivity is determined on the lower leg. The setup consists of a pneumatic tourniquet cuff, a computerized compressor and an electronic 10 cm Visual Analogue Scale (VAS). Double-Chambered Textile Tourniquet Cuffs (VBM Medizintechnik GmbH, Sulz, Germany) is used for pressure application.
  Measurements is carried out with the patient in supine position, and on the patient's dominant side. At all measurements a compression rate of 1.0kPa/sec is used. To minimize bias due to summation of pain, all measurements is carried out with a time interval of 5 minutes (the stimulus is repeated three times). Pain Threshold is defined as the pressure of the cuff at the subject's first sensation of pain when applying a constantly raising pressure (Unit kPa). Pain tolerance is defined as the pressure of the cuff when the pressure is switched off by the patient due to worst tolerable pain caused by pressure stimulation (Unit kPa).

CONTACTS AND LOCATIONS:
Locations (1):
- Esbjerg Hospital, Esbjerg, Denmark

IPD SHARING:
Plan to Share IPD: No